CLINICAL TRIAL: NCT06725277
Title: Comparative Effectiveness of Racemic Ketamine Versus Esketamine (Spravato®) for Depression: The OBSERVE Protocol
Brief Title: The OBSERVE Protocol
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2000038673; 23-005287 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Major Depression Disorder
MeSH Terms: interventions — Esketamine; Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IV Ketamine: Patients taking IV ketamine
  Interventions: Drug: IV Ketamine
- Spravato: Patients taking Spravato, an intranasal form of ketamine
  Interventions: Drug: Spravato

INTERVENTIONS:
Drug: Spravato — Intranasal esketamine
  Groups: Spravato
Drug: IV Ketamine — IV ketamine
  Groups: IV Ketamine

SUMMARY:
This observational protocol is intended to provide long-term follow-up data on patients initiating or continuing treatment with either Spravato® or IV ketamine. This can provide us information on the patient acceptability and satisfaction, patterns of use, long-term effectiveness, and safety of the two approaches.

This 5-year, 6-site study will enroll 450 total patients. The sites will comprise 3 academic medical centers and 3 community psychiatric practices.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet the following criteria:

1. Recently started treatment (within 75 days of screening visit) with IV ketamine or Spravato® as prescribed by a clinician for the treatment of moderate to severe (based on an initial MADRS score ≥ 25) TRD (refractory to two or more antidepressant trials) without psychotic features and having appropriate baseline measures collected before starting treatment. These patients are referred to as treatment-continuing subjects.

   OR
2. Scheduled to receive standard clinical treatment with IV ketamine or Spravato® as prescribed by a clinician for the treatment of moderate to severe (based on an initial MADRS score ≥ 25) TRD (refractory to two or more antidepressant trials) without psychotic features. These patients are referred to as treatment-initiating subjects.

   In addition, in order to be eligible, an individual must meet all of the following additional criteria:
3. Adult ages 18 or older
4. Provision of signed and dated informed consent form prior to any study procedures
5. Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Diagnosis of bipolar disorder or psychotic disorder (i.e., schizophrenia, schizoaffective disorder)
2. Other psychiatric comorbidities are permitted so long as depression is the predominant diagnosis
3. Active or recent (within 12 months) substance use disorder (other than nicotine)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population includes adults ages 18 or older with a diagnosis of major depressive disorder that is refractory to two or more antidepressant trials that have moderate to severe depression based on an initial MADRS score of 25 or greater having recently initiated treatment with appropriate baseline measures obtained (treatment-continuing) or scheduled to initiate standard clinical care (treatment-initiating) with either IV ketamine or Spravato® treatment.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-01-21 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
TSQM-9 | baseline to 6 months
  9-Item Treatment Satisfaction Questionnaire for Medication (TSQM-9). Analyses will be done for the whole sample as well as for treatment-continuing patients who recently completed a randomized trial of ketamine v. esketamine (EQUIVALENCE). The primary analysis for this measure will analyze treatment-continuing patients. Scores range from 0 - 100 with higher scores indicating higher satisfaction.

SECONDARY OUTCOMES:
Depression Severity (Self Report) | baseline to 6 months
  Change in 16-Item Quick Inventory of Depressive Symptomatology (QIDS). Score ranges from 0 - 27, with higher scores indicating worse depression.
Depression Severity (Clinician Report) | baseline to 6 months
  Change in Montgomery-Åsberg Depression Rating Scale (MADRS). Scores range from 0 - 60, with higher scores indicating worse depression.
Measure of Treatment Patterns: Number of treatments | baseline to 6 months
  Total number of treatments (ketamine or esketamine) during the study
Measure of Treatment Patterns: Reasons for Discontinuation | baseline to 6 months
  Number and proportion of patients who discontinue treatment
Measure of Treatment Patterns: Average Dose | baseline to 6 months
  Descriptive measures of average dose of ketamine / esketamine
Measures of Adverse Events | Baseline to 6 months
  Total number of serious adverse events possibly related to IV ketamine or esketamine

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Wilkinson, MD, Principal Investigator — Yale University
Locations (6):
- United States (6):
  - Mood Institute, Milford, Connecticut
  - Yale School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - LifeStance Health, Moore, Oklahoma
  - Houston Center for Advanced Psychiatric Treatment, Bellaire, Texas

IPD SHARING:
Plan to Share IPD: No